CLINICAL TRIAL: NCT02108093
Title: The Effect on Cerebral Oxygenation of Retrograde Autologous Priming of the Cardiopulmonary Bypass Circuit in Cardiac Surgery Patients: a Randomized Controlled Trial
Brief Title: The Effect on Cerebral Oxygenation of Retrograde Autologous Priming of the Cardiopulmonary Bypass Circuit in Cardiac Surgery Patients
Acronym: RAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amphia Hospital (Other)
Responsible Party: Principal Investigator, Thierry V Scohy, MD, PhD, Amphia Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAP
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RAP (retrograde autologous priming) group (Experimental): In the RAP (retrograde autologous priming) group, the priming solution is partially replaced by the patient's own circulating blood, before initiation of CPB. After initiation of cardiopulmonary bypass the priming volume is approximately 900 ml.
  Interventions: Procedure: retrograde autologous priming
- Control group (No Intervention): In the control group, the priming volume of the arterial and venous line will not be replaced by patient's own blood. The priming volume of cardiopulmonary bypass is 1300 ml in the control group.

INTERVENTIONS:
Procedure: retrograde autologous priming — Retrograde autologous priming (RAP) is a technique where, the patient's own circulating blood partially replaces the priming solution in the CPB.
  Other Names: RAP
  Arms: RAP (retrograde autologous priming) group

SUMMARY:
The effect of retrograde autologous priming (RAP) on regional cerebral oxygenation (rSO2) still remains unclear, because studies are limited in sample size and study design, and because of the absence of prospective studies. The investigators hypothesize that RAP limits the degree of hemodilution and thereby limits prolonged intraoperative cerebral desaturation during cardiopulmonary bypass (CPB), compared to the conventional priming method.

The primary objective of this study is to determine whether RAP limits the degree of hemodilution and limits prolonged intraoperative cerebral desaturation during cardiopulmonary bypass, compared to the conventional priming method. Prolonged intraoperative cerebral desaturation will be assessed by rSO2 desaturation score50. rSO2 desaturation score50 > 3000 is associated with increased risk of cognitive decline. The investigators hypothesize that RAP limits the degree of hemodilution and thereby limits the incidence of rSO2 desaturation score50 > 3000 with a relative difference of 50%.

The subjects who are divided in the RAP group, the retrograde autologous priming technique will be used, where the patient's own circulating blood partially will be replaced by the priming solution in the cardiopulmonary bypass. In the Control group the conventional priming method will be used. The main study parameters is rSO2 desaturation score50.

ELIGIBILITY:
Inclusion Criteria:

* Elective combined cardiac surgical procedures

Exclusion Criteria:

* Elective single cardiac surgical procedures
* off-pump procedure
* re-operation
* emergency operation
* methylene blue administration

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
prolonged intraoperative cerebral desaturation | Participants will be followed for the duration of the operation period, an expected average of 3 hours
  The primary study parameter of this study is prolonged intraoperative cerebral desaturation and will be assessed by rSO2 desaturation score50. rSO2 desaturation score50 > 3000 is associated with increased risk of cognitive decline. Formula described by Slater et al. : rSO2 score = 50% rSO2 - current rSO2 (%) x time (s) will be used to calculate the rSO2 score; from the intraoperative cerebral oximetry data.

SECONDARY OUTCOMES:
cerebral oxygenation desaturation episodes (CODE) | participants will be followed for the duriation of the operation period, an expected average of 3 hours
  CODE will be defined by a reduction of 20% baseline value of rSO2 at least one minute or an absolute reduction of 50%
Subjective Cognitive Failure Questionnaire (CFQ) | 3 months and 6 months after randomization
  Three and six months after randomization the Subjective CFQ will be sent to the patients to evaluate cognition.
blood transfusions (amount) | participants will be followed for the duration of ICU stay, an expected average of 2 days/ And participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  The amount of red blood cell transfusions the patient receive pre, peri and postoperatively during their stay in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Scohy, MD, PhD, Principal Investigator — Amphia Hospital
Locations (1):
- Amphia Hospital, Breda, Netherlands

REFERENCES:
- [Background] Slater JP, Guarino T, Stack J, Vinod K, Bustami RT, Brown JM 3rd, Rodriguez AL, Magovern CJ, Zaubler T, Freundlich K, Parr GV. Cerebral oxygen desaturation predicts cognitive decline and longer hospital stay after cardiac surgery. Ann Thorac Surg. 2009 Jan;87(1):36-44; discussion 44-5. doi: 10.1016/j.athoracsur.2008.08.070. PMID 19101265
- [Background] de Tournay-Jette E, Dupuis G, Bherer L, Deschamps A, Cartier R, Denault A. The relationship between cerebral oxygen saturation changes and postoperative cognitive dysfunction in elderly patients after coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):95-104. doi: 10.1053/j.jvca.2010.03.019. Epub 2010 Jul 22. PMID 20650659
- [Background] Murkin JM. Pathophysiological basis of CNS injury in cardiac surgical patients: detection and prevention. Perfusion. 2006 Jul;21(4):203-8. doi: 10.1191/0267659106pf869oa. PMID 16939113
- [Background] Hwang J, Huh J, Kim J, Park S, Hwang J, Nahm FS, Hahn S. The effect of retrograde autologous priming of the cardiopulmonary bypass circuit on cerebral oxygenation. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):995-9. doi: 10.1053/j.jvca.2011.02.017. Epub 2011 May 14. PMID 21576024
- [Background] Anastasiadis K, Argiriadou H, Kosmidis MH, Megari K, Antonitsis P, Thomaidou E, Aretouli E, Papakonstantinou C. Neurocognitive outcome after coronary artery bypass surgery using minimal versus conventional extracorporeal circulation: a randomised controlled pilot study. Heart. 2011 Jul;97(13):1082-8. doi: 10.1136/hrt.2010.218610. Epub 2011 Feb 28. PMID 21357641